CLINICAL TRIAL: NCT03465488
Title: Validation of Both Automated Quality Assured Egg Counting System and Molecular Markers for Monitoring the Spread of Anthelmintic Resistance.
Brief Title: Validating Egg-based Diagnostics and Molecular Markers for the Spread of Anthelmintic Resistance
Acronym: StarwormsWP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other)
Responsible Party: Principal Investigator, Virologie, Professor, University Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPP1120972
Record Dates: First submitted 2018-02-16; First posted 2018-03-14 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Soil-transmitted Helminth Infections
Keywords: parasitology; helminth infections; diagnosis; drug resistance; albendazole; benzimidazole drugs; Ascaris; Trichuris; hookworm; qPCR; microscopy
MeSH Terms: conditions — Trematode Infections; Disease; Ancylostomiasis | interventions — Albendazole; halofantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects (Experimental): All participants that meet all inclusion criteria and none of the exclusion criteria will be enrolled in the study and receive a subject identifier (SubjectID). At baseline, all participants will receive a single treatment of albendazole 400mg and their stool will be examined for helminth eggs. Two to three weeks after treatment a follow-up examination of their stool is performed.
  Interventions: Drug: Albendazole Pill 400mg (GSK)

INTERVENTIONS:
Drug: Albendazole Pill 400mg (GSK) — One single dose of 400mg Albendazole is provided at baseline.
  Other Names: Albendazole 400mg form GlaxoSmithKline (Batch Nr: 335726)

SUMMARY:
Soil-transmitted helminths (STHs) are a group of parasitic worms that infect millions of children in sub-tropical and tropical countries, resulting in malnutrition, growth stunting, intellectual retardation and cognitive deficits. To control the morbidity due to these worms, school-based deworming programs are implemented, in which anthelminthic drugs are administered to children without prior diagnosis. The continued fight against these worms is aided by the London declaration on neglected tropical diseases, which helps sustain and expand global drug donation program, resulting in an unprecedented growth of deworming programs. However, the high degree of drug pressure makes deworming programs vulnerable to the development of anthelmintic resistance because they only rely on one drug with sometimes suboptimal efficacy and there is no availability of alternative drugs. Moreover, at present, there is no surveillance system to monitor the emergence and spread of anthelmintic resistance. It remains unclear to what extent the efficacy of drugs may have dropped and whether anthelmintic resistance is already present.

This project aims to strengthen the monitoring and surveillance of drug efficacy and anthelmintic resistance in STH programs. As such, it will support deworming programs in their quest to eliminate STHs as a public health problem.

The specific objectives of the first work package are to validate diagnostic tools to monitor drug efficacy and the spread of anthelmintic resistance, and to validate molecular markers for benzimidazole resistance.

This study will be conducted at four different sites (Ethiopia, Tanzania, Lao PDR and Brazil) and will focus on school-aged children (age 5-14). At baseline subjects will be asked to provide a recent stool sample which will be processed using 3 different microscopic techniques (KK, Mini-Flotac and FECPAKG2). All children will be treated with a single-oral dose of albendazole (ALB) 400 mg and 14-21 days after treatment, a second stool sample will be collected from all children to again determine the fecal egg counts. At each sampling, stool is stored in preservative. Stored stool will be shipped to Belgium for DNA extraction and quantitative PCR (qPCR) analysis. A subset of the samples will be analysed by pyrosequencing to evaluate the single nucleotide polymorphisms in the b-tubulin gene. Pooling of the stored samples will also be performed to compare with the values obtained from analysing individual samples.

DETAILED DESCRIPTION:
Background Soil-transmitted helminths (STHs) are a group of parasitic worms that infect millions of children in sub-tropical and tropical countries, resulting in malnutrition, growth stunting, intellectual retardation and cognitive deficits. To control the morbidity due to these worms, school-based deworming programs are implemented, in which anthelminthic drugs are administered to children without prior diagnosis. The continued fight against these worms is aided by the London Declaration on Neglected Tropical Diseases, which helps sustain and expand global drug donation program, resulting in an unprecedented growth of deworming programs. to illustrate, in the last four years the coverage of mass drug administration (MDA) has doubled from 30 to 60%, and ongoing global efforts are made to ultimately reach the milestone of 75% by 2020.

Threats While the laudable long-term aim is to eliminate STHs as a public health problem by 2020, and to eventually declare targeted geographical areas free from infections, this high degree of drug pressure makes deworming programs vulnerable to the development of anthelmintic resistance because the programs only rely on one drug with sometimes suboptimal efficacy and there is no availability of alternative drugs.

Challenges

At present, there is no surveillance system to monitor the emergence and spread of anthelmintic resistance. It remains unclear to what extent the efficacy of drugs may have dropped and whether anthelmintic resistance is already present. However, developing such a system is not straightforward. Deworming programs typically operate in resource-constrained settings, and program managers require some flexibility to minimize both financial and technical resources, while ensuring a reliable assessment of the drug efficacy. The most important obstacles to globally monitor patterns of changing drug efficacy and spread of anthelmintic resistance are the following:

* the shortage of diagnostic laboratories with experienced staff to perform the surveys and analyze and report the obtained data
* the absence of a quality assurance system that guarantees auditable results
* the lack of guidance in designing surveys as the programs progresses
* the lack of data supporting the validity of molecular markers to detect anthelmintic resistance in human STHs
* the lack of sensitive and point-of-care tools that allow the detection of low frequencies of anthelmintic resistance Main objective This project aims to strengthen the monitoring and surveillance of drug efficacy and anthelmintic resistance in STH programs. As such, it will support deworming programs in their quest to eliminate STHs as a public health problem by 2020.

The specific objectives of the first part of the project are to validate diagnostic tools to monitor drug efficacy and the spread of anthelmintic resistance, and to validate molecular markers for benzimidazole resistance.

Study protocol This study will conducted at four different sites at Africa (Ethiopia and Tanzania), Asia (Lao PDR) and Latin-America (Brazil). The selection of these sites is based on their experience in assessing drug efficacy and evaluating the performance of diagnostic tools, the availability of well-equipped diagnostic facilities and skilled personnel, and their national MDA history.

The study will focus on school-aged children (age of 5 to 14 years). At baseline subjects will be asked to provide a recent (within 4 hours) stool sample of at least 9 grams. All stool samples will be processed using the FECPAKG2, a duplicate Kato-Katz thick smear (the most commonly applied fecal egg count (FEC) technique) and Mini-Flotac (a novel technique that has a sensitivity at least equal to that of Kato-Katz). All children providing a stool sample will be provided a single-oral dose of ALB 400 mg under supervision. Fourteen to 21 days after treatment, a second stool sample will be collected from all the children that proved positive for any STH species at baseline to determine the FECs.

At each sampling, 2x 1 gram of stool is stored in preservative for downstream molecular analysis. Stored stool will be shipped to Belgium for DNA extraction and qPCR analysis. A subset of the samples will be analysed by Pyrosequencing to evaluate the single nucleotide polymorphisms in the b-tubulin gene.

Pooling of the stored samples will also be performed to compare with the values obtained from analysing individual samples.

Data handling Data will first be recorded on specific study record forms. These results will then be entered into the custom designed Excel-files by two different data entry clerks to minimize errors in data due to incorrect data entry.

Study management Studies in the different sites will be organized and supported out of Ghent University. The project team members will travel to each individual trial site to train local personnel in the different coprological techniques and to get them acquainted with the trial protocol and documents.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, is 5-14 years of age
* Subject is otherwise in an healthy condition (medical history and physical examination)
* Parent(s)/guardians of subjects (or their legally-accepted representatives) signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to have their child participate in the study.
* Subject of ≥6 years has assented (agreed) to participate in the study.
* Subject of ≥12 has signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* The subject swallowed the entire drug (ALB 400 mg) under supervision
* Subject provides a stool sample of at least 9 grams

Exclusion Criteria:

* Subject has active diarrhea (defined as the passage of 3 or more loose or liquid stools per day) at baseline or follow-up
* Subject has any acute medical condition or is experiencing a severe concurrent medical condition
* Subject has a known hypersensitivity to benzimidazole drugs
* Subject has received an anthelminthic treatment within 90 of the start of the treatment.
* Subject vomited within 4 hours after drug administration
* Subject is unable to provide a stool sample at follow-up

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Validation of the performance of FECPAKG2 to assess drug efficacy | up to 12 months
  We will validate the performance of the FECPAKG2 as well as its ability to assess drug efficacy by means of egg reduction rates.
In depth evaluation of the FECPAKG2 technique to assess drug efficacy | up to 12 months
  We will check the variation in egg counts obtained in repeated measurements and by different technicians and make a cost assessment.
Validation of b-tubulin gene as a molecular marker for benzimidazole resistance | up to 24 months
  This will be done through assessment of the polymorphisms at the b-tubulin gene using a pyrosequencing approach. We will compare results obtained from the 4 different study sites which have a varying MDA history as well as results obtained from responders, poor responders and non-responders within each different site.

SECONDARY OUTCOMES:
Comparing the sensitivity of quantitative PCR with traditional diagnostic tools (Kato-Katz, Mini-FLOTAC and FECPAKG2) for the detection of soil-transmitted helminth infections. | up to 12 months
  It is commonly accepted that molecular tools are more sensitive to traditional diagnostic tools, however studies comparing qPCR with a wide range of traditional microscopic techniques are scarce. In this project we will evaluate the performance of qPCR in terms of sensitivity to detect infection compared to the results obtained by coprological analysis of samples by Kato-Katz, Mini-FLOTAC and FECPAKG2.
Comparing the use of individual and pooled stool samples to assess polymorphisms in the β-tubulin gene. | up to 24 months
  Pyrosequencing results for β-tubulin gene from individual samples will be compared to those from pooled samples. This will shed a light on whether or not pooling stool samples provides similar information regarding the presence of single nucleotide polymorphisms as when compared to evaluating individual samples. This is important because pooling samples would allow important cuts in both technical and financial resources to process the samples.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Levecke, PhD, Principal Investigator — University Ghent
Locations (4):
- Fiocruz - Research institute of Renê Rachou, Belo Horizonte, Minas Gerais, Brazil
- Jimma University, Jimma, Ethiopia
- National Institute of Public Health, Vientiane, Laos
- The Public Health Laboratory - Ivo de Carneri (PHL-IdC), Chake Chake, Pemba, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
De-identified results will be shared online and with collaborating researchers for further extensive analysis.
Supporting Information: Study Protocol, SAP
Time Frame: A general overview of the project is already published on our project website. The specific study protocol for work-package 1 of the project is currently being submitted for publication. Once final data is collected, De-identified data will be available through the project website as well. No specific time-frame will be applied.
Access Criteria: Free access for all
URL: https://www.starworms.org/tools/overview/starworms-documents

REFERENCES:
- [Derived] Coffeng LE, Vlaminck J, Cools P, Denwood M, Albonico M, Ame SM, Ayana M, Dana D, Cringoli G, de Vlas SJ, Fenwick A, French M, Kazienga A, Keiser J, Knopp S, Leta G, Matoso LF, Maurelli MP, Montresor A, Mirams G, Mekonnen Z, Correa-Oliveira R, Pinto SA, Rinaldi L, Sayasone S, Steinmann P, Thomas E, Vercruysse J, Levecke B. A general framework to support cost-efficient fecal egg count methods and study design choices for large-scale STH deworming programs-monitoring of therapeutic drug efficacy as a case study. PLoS Negl Trop Dis. 2023 May 17;17(5):e0011071. doi: 10.1371/journal.pntd.0011071. eCollection 2023 May. PMID 37196017
- [Derived] Walker M, Cools P, Albonico M, Ame SM, Ayana M, Dana D, Keiser J, Matoso LF, Montresor A, Mekonnen Z, Correa-Oliveira R, Pinto SA, Sayasone S, Vercruysse J, Vlaminck J, Levecke B. Individual responses to a single oral dose of albendazole indicate reduced efficacy against soil-transmitted helminths in an area with high drug pressure. PLoS Negl Trop Dis. 2021 Oct 19;15(10):e0009888. doi: 10.1371/journal.pntd.0009888. eCollection 2021 Oct. PMID 34665810
- [Derived] Vlaminck J, Cools P, Albonico M, Ame S, Ayana M, Cringoli G, Dana D, Keiser J, Maurelli MP, Matoso LF, Montresor A, Mekonnen Z, Mirams G, Correa-Oliveira R, Pinto SA, Rinaldi L, Sayasone S, Thomas E, Vercruysse J, Verweij JJ, Levecke B. Therapeutic efficacy of albendazole against soil-transmitted helminthiasis in children measured by five diagnostic methods. PLoS Negl Trop Dis. 2019 Aug 1;13(8):e0007471. doi: 10.1371/journal.pntd.0007471. eCollection 2019 Aug. PMID 31369562
- [Derived] Cools P, Vlaminck J, Albonico M, Ame S, Ayana M, Jose Antonio BP, Cringoli G, Dana D, Keiser J, Maurelli MP, Maya C, Matoso LF, Montresor A, Mekonnen Z, Mirams G, Correa-Oliveira R, Pinto SA, Rinaldi L, Sayasone S, Thomas E, Verweij JJ, Vercruysse J, Levecke B. Diagnostic performance of a single and duplicate Kato-Katz, Mini-FLOTAC, FECPAKG2 and qPCR for the detection and quantification of soil-transmitted helminths in three endemic countries. PLoS Negl Trop Dis. 2019 Aug 1;13(8):e0007446. doi: 10.1371/journal.pntd.0007446. eCollection 2019 Aug. PMID 31369558
- [Derived] Vlaminck J, Cools P, Albonico M, Ame S, Ayana M, Bethony J, Cringoli G, Dana D, Keiser J, Maurelli MP, Montresor A, Mekonnen Z, Mirams G, Correa-Oliveira R, Prichard R, Rashwan N, Rinaldi L, Sayasone S, Thomas E, Verweij JJ, Vercruysse J, Levecke B. Comprehensive evaluation of stool-based diagnostic methods and benzimidazole resistance markers to assess drug efficacy and detect the emergence of anthelmintic resistance: A Starworms study protocol. PLoS Negl Trop Dis. 2018 Nov 2;12(11):e0006912. doi: 10.1371/journal.pntd.0006912. eCollection 2018 Nov. PMID 30388108
- See also: Project website — https://www.starworms.org
- See also: Laboratory website — http://www.vetparasitology.ugent.be/